CLINICAL TRIAL: NCT01201538
Title: A Phase II Study of Nilotinib in Growing Vestibular Schwannomas
Brief Title: A Study of Nilotinib in Growing Vestibular Schwannomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study PI passed away We had trouble recruiting for the drug arm
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-024
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Growing Vestibular Schwannomas
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
Acoustic Neuromas (otherwise known as Vestibular Schwannoma -VS) are benign tumors which grow on the hearing nerve and can cause progressive hearing loss and compression of vital brain structures and even death if it continues. The primary objective of this study is to evaluate the efficacy of Nilotinib in the treatment of patients with progressing VS. Secondary objectives of this study is to evaluate the toxicity profile, quality of life and symptom management of Nilotinib in the treatment of patients with progressing VS.

DETAILED DESCRIPTION:
UHN laboratory has demonstrated that targets of Imatinib (c-Kit and PDGFR-α and PDGFR-ß) are overexpressed and activated in both sporadic and NF2 VS.It has also been shown pre-clinically that Imatinib induced a reduction in proliferation and cell viability, with increased apoptosis, in HEI-193 human NF2-null VS cells.Nilotinib is a newer generation RTK inhibitor, with a similar target profile as Imatinib. It was designed by modifying the Imatinib molecule62, and has 30-fold increased potency compared to IImatinib43. In clinical studies of patients with CML or GIST resistant to Imatinib, Nilotinib has demonstrated efficacy with minimal toxicity. Nilotinib (Tasigna®, code number AMN107) was first approved in 2007 for use in Philadelphia chromosome positive CML in the chronic or accelerated phase in patients resistant or intolerant to prior therapy. Thus making Nilotinib an ideal drug to study in understanding its benefit in VS patients.

ELIGIBILITY:
Inclusion

1. Age >18 years of age with either sporadic or NF-2 associated VS
2. Growing VS defined as an increase in MRI volumetric growth (minimal 15%) on two successive scans within 18 months prior to registration
3. Patients may be either treatment naïve or have recurrent VS after previous surgery/ stereotactic radiosurgery
4. Essentially neurologically asymptomatic (with the exception of sensorineural hearing loss, mild tinnitus and facial numbness) as assessed by the investigator
5. Karnofsky performance score >70
6. Adequate renal, haematological, liver function within 7 days prior to registration
7. Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions
8. Willingness and ability to provide informed consent

Exclusion

1. Brain stem compression with symptoms
2. Symptomatic hydrocephalus
3. T2/Flair signal changes with distortion of adjacent brain stem and IVth ventricle
4. Lower cranial nerve dysfunction
5. Concurrent or previous invasive malignancy, except adequately treated non-melanoma skin cancer or other solid tumours curatively treated with no evidence of disease for ≥ 3 years
6. Evidence of severe or uncontrolled systemic disease which in the opinion of the investigator makes it undesirable for the subject to participate in the study
7. Known hypersensitivity to the study drug or drug of similar chemical or biological composition
8. Impaired cardiac function including

   1. Congenital long QT syndrome or family history of long QT syndrome
   2. Clinically significant resting bradycardia (< 50 beats per minute)
   3. Myocardial infarction within 1 year prior to registration or other clinically significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)
   4. History of or current clinically significant ventricular or atrial tachyarrhythmia
   5. QTcF > 450 msec on screening ECG. If QTcF > 450 msec and electrolytes are not within normal ranges then electrolytes should be corrected and the patient rescreened for QTcF.
   6. Unable to monitor the QT/QTc interval on ECG
9. Treatment with strong CYP3A4 inhibitors or CYP3A4 inducers and treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
10. Treatment with any medications that have the potential to prolong the QT interval and cannot be either discontinued or switched to a different medication prior to starting study drug.
11. Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug
12. History of acute or pancreatic disease within one year of study registration or past medical history of chronic pancreatitis.
13. Acute liver disease
14. History of significant congenital or acquired bleeding disorder
15. Use of any investigational agent within 28 days prior to enrollment in the study or foreseen use of an investigational agent during the study
16. Women who are pregnant or breastfeeding or of childbearing potential without a negative serum pregnancy test within 7 days prior to registration. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male or female patients of childbearing potential unwilling to use effective barrier contraceptives or medical contraceptive to avoid pregnancy throughout the trial and for 3 months following discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
volume change of Vestibular Schwannoma | 3 years - 1 year drug treatment, 2 year follow-up
  Primary Outcomes of interest will be volumetric tumor response and lack of tumor progression. A response to treatment will be defined as a 20% or greater, change in volume, as defined by Plotkin et al.

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Guha, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario